CLINICAL TRIAL: NCT01215994
Title: Comparative Study of New Formulae of GFR Estimation Based on Creatinine, Cystatin C and Cr51-EDTA.
Brief Title: Estimation of Glomerular Filtration Rate (GFR) in Patients With Type 2 Diabetes Mellitus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Fotios Iliadis, MD, ASSISTANT PROFESSOR, AHEPA University Hospital
Other Study IDs: AHEPA
Record Dates: First submitted 2010-08-30; First posted 2010-10-07 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the present study is to evaluate bias, precision and accuracy of new cystatin C and creatinine based equations for GFR estimation compared with 51Cr-EDTA (chromium-51 labeled ethylenediamine tetraacetic acid) measured GFR in patients with diabetes.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate bias, precision and accuracy of new cystatin C and creatinine based equations for GFR estimation compared with 51Cr-EDTA measured GFR in patients with diabetes.

Additional, we will check which equation detects better the reduction of renal function over the time, in patients with diabetes.

Finally, we will investigate if cystatin C levels can be influenced by factors other than GFR

ELIGIBILITY:
Inclusion Criteria:

* Type 2 and type 1 diabetes mellitus

Exclusion Criteria:

* Patients with other type diabetes: gestational, exocrine pancreatic defects, endocrinopathies, drugs
* Patients with end-stage renal disease, cardiac failure, hepatic failure, malignancies, immunosuppression, pregnant, diabetic ketoacidosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients treated in the primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Grekas, PhD, MD, Study Chair — Aristotle University of Thessaloniki, Greece
Locations (1):
- AHEPA University Hospital of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Iliadis F, Didangelos T, Ntemka A, Makedou A, Moralidis E, Gotzamani-Psarakou A, Kouloukourgiotou T, Grekas D. Glomerular filtration rate estimation in patients with type 2 diabetes: creatinine- or cystatin C-based equations? Diabetologia. 2011 Dec;54(12):2987-94. doi: 10.1007/s00125-011-2307-1. Epub 2011 Sep 23. PMID 21947381